CLINICAL TRIAL: NCT01425463
Title: A Double-blind, Double-dummy, Parallel, Active-controlled, Randomized and Multi-center Trial to Investigate Efficacy and Safety in Subjects With Iron Deficiency Anemia for Ferrous (II) Glycine Sulphate Complex Versus Polyferose Capsules Therapy
Brief Title: A Double-blind, Double-dummy, Parallel, Active-controlled, Randomized Trial to Evaluate Efficacy & Safety in Anemia Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanol GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0986; 2014-004380-20 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Ferrous (II) Glycine Sulphate Complex; Polyferose; Ferro Sanol duodenal; Niferex; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferroglycine sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous (II) Glycine Sulphate Complex (Experimental): Ferrous (II) Glycine Sulphate Complex treatment with 567.7 mg three times a day (t.i.d.) for 12 weeks plus Placebo to Polyferose.
  Interventions: Drug: Ferrous (II) Glycine Sulphate Complex; Other: Placebo to Polyferose
- Polyferose (Active Comparator): Polyferose treatment with 150 mg twice daily (b.i.d) for 12 weeks plus Placebo to Ferrous (II) Glycine Sulphate Complex.
  Interventions: Drug: Polyferose; Other: Placebo to Ferrous (II) Glycine Sulphate Complex

INTERVENTIONS:
Drug: Ferrous (II) Glycine Sulphate Complex — Oral dose of 567.7 mg Ferrous (II) Glycine Sulphate Complex three times a day (t.i.d) for 12 weeks (equivalent to 300 mg iron element per day for 12 weeks).
  Administered orally with water.
  Other Names: Ferro Sanol Duodenal
  Arms: Ferrous (II) Glycine Sulphate Complex
Drug: Polyferose — Oral dose of 150 mg Polyferose Capsules twice daily (b.i.d) for 12 weeks (equivalent to 300 mg iron element per day for 12 weeks).
  Administered orally with water.
  Other Names: Nifirex
  Arms: Polyferose
Other: Placebo to Ferrous (II) Glycine Sulphate Complex — Administered orally with water.
  Arms: Polyferose
Other: Placebo to Polyferose — Administered orally with water.
  Arms: Ferrous (II) Glycine Sulphate Complex

SUMMARY:
To evaluate the efficacy and safety of 12 weeks treatment with Ferrous (II) Glycine Sulphate Complex in comparison to Polyferose capsules in Chinese subjects with manifest Iron Deficiency Anemia.

ELIGIBILITY:
Inclusion Criteria:

* An iron deficiency anemia patient with Serum Ferritin < 12 ng/mL, serum Hb-values >60 and < 120 g/L in males, < 110 g/L in females

Exclusion Criteria:

* With any Mal-absorption Syndrome
* With a history of Thalassemia or Sickle Cell Anemia
* With untreated concurrent Vitamin B12 or Folate deficiency at Baseline

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (15):
- China (15):
  - 15, Changsha
  - 16, Changsha
  - 1, Fuzhou
  - 10, Guangzhou
  - 5, Hangzhou
  - 6, Hangzhou
  - 7, Jinan
  - 8, Jinan
  - 13, Shanxi
  - 14, Shanxi
  - 12, Shenyang
  - 2, Tianjin
  - 17, Wenzhou
  - 4, Wuxi
  - 9, Xi'an

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in March 2011 in order to end up with 16 centers in China with enrolled subjects.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS). The RS includes all subjects who have a randomization number recorded on the Case Report Form (CRF).
Groups:
- Ferrous (II) Glycine Sulphate Complex: Ferrous (II) Glycine Sulphate Complex treatment with 567.7 mg three times a day (t.i.d.) for 12 weeks plus Placebo to Polyferose.
  Ferrous (II) Glycine Sulphate Complex: Oral dose of 567.7 mg Ferrous (II) Glycine Sulphate Complex three times a day (t.i.d) for 12 weeks (equivalent to 300 mg iron element per day for 12 weeks).
  Administered orally with water.
  Placebo to Polyferose: Administered orally with water.
- Polyferose: Polyferose treatment with 150 mg twice daily (b.i.d) for 12 weeks plus Placebo to Ferrous (II) Glycine Sulphate Complex.
  Polyferose: Oral dose of 150 mg Polyferose Capsules twice daily (b.i.d) for 12 weeks (equivalent to 300 mg iron element per day for 12 weeks).
  Administered orally with water.
  Placebo to Ferrous (II) Glycine Sulphate Complex: Administered orally with water.
Period: Overall Study
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Started | 130 | 126
Safety Set | 126 | 122
Full Analysis Set | 122 | 116
Completed | 106 | 102
Not Completed | 24 | 24
Not completed — Adverse Event | 5 | 7
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Unknown Reason | 4 | 7

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Full Analysis Set (FAS). FAS consists of all enrolled subjects who took at least one dose of study medicine and have at least one post-baseline effectiveness measurement (Hemoglobin-value). It also includes subjects with protocol deviance and incomplete data due to withdrawal.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose | Total
Number analyzed (Participants) | 122 | 116 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (8.5) | 37.8 (7.9) | 37.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 115 | 237
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 122 | 116 | 238
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 122 | 116 | 238
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 58.2 (7.8) | 58.1 (7.6) | 58.1 (7.7)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 161.2 (4.4) | 161.2 (4.6) | 161.2 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) From Baseline (Week 0) to Week 12
Time Frame: From Baseline to Week 12
Population: The Analysis Population refers to the Per-Protocol Set (PPS), which is defined as a subset of the FAS, excluding all subjects with protocol deviations considered important for the subjects' validity concerning the efficacy analysis.
Measure: Mean (Standard Deviation); unit: gramm per liter (g/L)
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Number analyzed (Participants) | 95 | 92
gramm per liter (g/L) | 31.47 (23.77) | 31.92 (21.82)
Statistical Analysis 1: Comparison: Ferrous (II) Glycine Sulphate Complex vs Polyferose; Test type: Non-Inferiority or Equivalence — Noninferiority of the investigational drug (Ferrous (II) Glycine Sulphate Complex) to the reference drug (Polyferose) was concluded if the lower limit of the two-sided 95 % confidence interval was greater than -7.0 g/L; LS-Mean of ANCOVA = -2.19, 95% CI 2-sided [-8.47 to 4.09]

2. Secondary Outcome: Change in Hemoglobin (Hb) From Baseline (Week 0) to Week 2
Time Frame: From Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gramm per liter (g/L)
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Number analyzed (Participants) | 93 | 91
gramm per liter (g/L) | 12.29 (13.60) | 12.79 (13.13)

3. Secondary Outcome: Change in Hemoglobin (Hb) From Baseline (Week 0) to Week 4
Time Frame: From Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gramm per liter (g/L)
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Number analyzed (Participants) | 95 | 92
gramm per liter (g/L) | 20.37 (19.63) | 20.16 (17.46)

4. Secondary Outcome: Change in Hemoglobin (Hb) From Baseline (Week 0) to Week 8
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gramm per liter (g/L)
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Number analyzed (Participants) | 95 | 92
gramm per liter (g/L) | 26.57 (22.67) | 28.33 (20.90)

5. Secondary Outcome: Percentage of Responders at Week 12
Description: Responders are defined as having an increment of Hemoglobin (Hb) > 15 g/L and post-treatment Hb > 120 g/L (male) or > 110 g/L (female) at Visit 6 (Week 12).
Time Frame: End of Treatment Period (Week 12)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Number analyzed (Participants) | 95 | 92
percentage of participants | 71.6 | 80.4

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 14 weeks from Baseline to the Safety Follow-Up Visit.
Description: Adverse Events refer to the Safety Set (SS). SS represents all subjects included in the study who took at least one dose of study medication and have at least one safety evaluation after that.
Arm/Group | Ferrous (II) Glycine Sulphate Complex | Polyferose
Serious Adverse Events (participants affected / at risk) | 3/126 | 3/122
Other Adverse Events (participants affected / at risk) | 22/126 | 25/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferrous (II) Glycine Sulphate Complex (N=126) | Polyferose (N=122)
Abortion induced (Surgical and medical procedures) | 2 (2) | 1 (1)
Measles (Infections and infestations) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferrous (II) Glycine Sulphate Complex (N=126) | Polyferose (N=122)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 11 (14)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 5 (6)
Melaena (Gastrointestinal disorders) | 6 (6) | 8 (9)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days